CLINICAL TRIAL: NCT06269107
Title: A 40-week Study Comparing the Efficacy and Safety of Once Weekly IcoSema and Daily Insulin Glargine 100 Units/mL in Participants With Type 2 Diabetes Inadequately Controlled on Oral Anti Diabetic Drugs COMBINE 4
Brief Title: A Research Study to See How Well New Weekly Medicine IcoSema, Which is a Combination of Insulin Icodec and Semaglutide, Controls Blood Sugar Levels in People With Type 2 Diabetes (T2D), Compared to Daily Insulin Glargine (COMBINE 4)
Acronym: COMBINE 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1535-4988; U1111-1283-8648 (Other: World Health Organization (WHO)); 2022-502484-38-00 (Other: European Medicines Agency (EMA))
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IcoSema (Experimental): Participants will receive once weekly IcoSema subcutaneously with or without oral anti diabetic drugs for 40 weeks.
  Interventions: Drug: IcoSema
- Insulin glargine (Experimental): Participants will receive once daily insulin glargine subcutaneously with or without oral anti diabetic drugs for 40 weeks.
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: IcoSema — IcoSema will be administered subcutaneously.
  Arms: IcoSema
Drug: Insulin glargine — Insulin glargine will be administered subcutaneously.
  Arms: Insulin glargine

SUMMARY:
This study will compare the new medicine IcoSema, which is a combination of insulin icodec and semaglutide, taken once a week, to insulin glargine (mentioned as insulin glargine in this form) taken daily in people with type 2 diabetes. The study will look at how well IcoSema controls blood sugar levels as compared to insulin glargine in people with type 2 diabetes who do not have their blood sugar properly controlled with other oral diabetes medicines. Participant will either get IcoSema or insulin glargine. Which treatment participants get is decided by chance. IcoSema is a new medicine that doctors cannot prescribe. Doctors can already prescribe insulin glargine in many countries. The study will last for about 11 months (47 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Male or female and age above or equal to 18 years at the time of signing the informed consent.
* Diagnosed with T2D greater than or equal to (≥) 180 days before screening.
* HbA1c ≥ 8.0% (≥ 64.0 millimoles per mole [mmol/mol]) as assessed by central laboratory on the day of screening.
* Insulin naïve. Short term insulin treatment for a maximum of 14 consecutive days before screening is allowed, as is prior insulin treatment for gestational diabetes.
* Currently treated with 1-3 oral anti diabetic drug (OADs) with stable daily doses ≥ 90 days before screening comprising any of the following anti diabetic drug(s) at effective or maximum tolerated dose.

  * Metformin
  * Sulfonylureas
  * Meglitinides (glinides)
  * Dipeptidyl peptidase (DPP) 4 inhibitors
  * Sodium glucose co transporter 2 inhibitors
  * Alpha glucosidase inhibitors
  * Thiazolidinediones
  * Marketed oral combination products only including the products listed above.
* Body mass index (BMI) less than or equal to (≤) 40.0 kilogram per square meter (kg/m^2).

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbaring potential and not using highly effective contraceptive method.
* Anticipated initiation or change in concomitant medication (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or systemic corticosteroids).
* Any episodes of diabetic ketoacidosis or treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening.
* Presence or history of pancreatitis (acute or chronic) within 180 days before screening.
* Any of the following: Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 180 days before screening.
* Chronic heart failure classified as being in New York Heart Association Class IV at screening.
* Recurrent severe hypoglycaemic episodes within the last year (12 months) as judged by the investigator.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days before screening or in the period between screening and randomisation. Pharmacological pupil dilation is a requirement unless using a digital fundus photography camera specified for non dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to week 40
  Measured in percentage (%)-point.

SECONDARY OUTCOMES:
Change in body weight | From baseline (week 0) to week 40
  Measured in kilogram (kg).
Time in range 3.9-10.0 millimoles per liter (mmol/L) (70-180 milligram per deciliter [mg/dL]) | From week 36 to week 40
  Measured in % of readings.
Time spent less than (<) 3.0 mmol/L (54 mg/dL) | From week 36 to week 40
  Measured in % of readings.
Time spent greater than (>) 10.0 mmol/L (180 mg/dL) | From week 36 to week 40
  Measured in % of readings.
Weekly basal insulin dose | From week 38 to week 40
  Measured in units of insulin.
Change in fasting plasma glucose (FPG) | From baseline (week 0) to week 40
  Measured in mmol/l.
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQs) in total treatment satisfaction | From baseline (week 0) to week 40
  The DTSQs items are scored on a 7-point graded response scale ranging from 0 to 6. Score ranges from 0 to 36. Higher scores indicate greater the satisfaction with medication.
Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by blood glucose meter) or severe hypoglycaemic episodes (level 3) | From baseline (week 0) to week 45
  Measured in number of episodes.
Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL), confirmed by BG meter) | From baseline (week 0) to week 45
  Measured in number of episodes.
Number of severe hypoglycaemic episodes (level 3) | From baseline (week 0) to week 45
  Measured in number of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (91):
- United States (29):
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - First Valley Med Grp Lancaster, Lancaster, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Clinical Trials Research_Sacramento, Sacramento, California
  - Northeast Research Institute, Fleming Island, Florida
  - Clinical Research of Cent FL, Winter Haven, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Endeavor Health, Skokie, Illinois
  - Cotton-O'Neil Diab & Endo Ctr, Topeka, Kansas
  - Methodist Phys. Clinic, Omaha, Nebraska
  - Albuquerque Clin Trials, Inc., Albuquerque, New Mexico
  - AMC Community Endocrinology, Albany, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Physician's East Endocrinology, Greenville, North Carolina
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Advanced Medical Research, Maumee, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Velocity Clinical Research- Cedar Park, Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Diabetes and Thyroid Ctr of FW, Fort Worth, Texas
  - Fmc Science, Llc, Lampasas, Texas
  - Quality Research Inc, San Antonio, Texas
  - Flourish Research, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - TPMG Clinical Research, Newport News, Virginia
- China (9):
  - Peking University People's Hospital-Endocrinology, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University-Endocrinology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Huizhou Central People's Hospital-Endocrinology, Huizhou, Guangdong
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Pudong New Area People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
- Greece (6):
  - Evangelismos Hospital, Athens
  - 'G. Gennimatas' General Hospital of Athens, Athens
  - "Laiko" General Hospital of Athens, Athens
  - General Hospital of Kalamata, Kalamata
  - Univ Gen Hospital Larisa, Larissa
  - "Thermi" Private Hosital, Thessaloniki
- India (11):
  - Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - BYL Nair Hospital and T N Medical College Department of endo, Mumbai, Maharashtra
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - BSES MG hospital, Mumbai, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Udyaan Health Care, Lucknow, Uttar Pradesh
  - Post Graduate Institute of Medical Education & Research, Chandigarh
- Italy (8):
  - ASL Avezzano Sulmona L'Aquila - Ospedale San Salvatore - UOC Diabetologia, L’Aquila, Abbruzzo
  - Casa Sollievo della Sofferenza reparto endocrinologia, San Giovanni Rotondo, FG
  - A.O.U. Policlinico Umberto I, Rome, Lazio
  - I.N.R.C.A. Istituto Nazionale di Riposo E Cura Per Gli Anziani, Ancona
  - Casa della Salute di Ceccano - Ambulatori Campus Biomedico, Ceccano (Frosinone)
  - ASL 4 Chiavarese, Chiavari (genova)
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera di Perugia;Ospedale S. Maria della Misericordia, Perugia
- Japan (7):
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - Tokuyama clinic_Diabetic internal medicine, Chiba
  - Oodouri Diabetes, Internal medicine Clinic_Internal Medicine, Diabetes Internal Medicine, Hokkaido
  - Oyama East Clinic_Internal Medicine, Tochigi
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Juntendo University Hospital, Tokyo
- Poland (10):
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok, Podlaskie Voivodeship
  - SNZOZ Lege Artis, Bialystok
  - Grazyna Pulka Specjalistyczny Osrodek "All-Med", Krakow
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Centrum Terapii Współczesnej J.M. Jasnorzewska S.K.A., Lodz
  - Velocity Nova Sp. z o.o., Lublin
  - NBR Polska Tomasz Klodawski, Warsaw
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw
  - Clinhouse Centrum Medyczne, Zabrze
  - Velocity Nova Sp. z o.o., Staszów, Świętokrzyskie Voivodeship
- Advanced Clinical Research LLC, Bayamón, Puerto Rico
- South Africa (6):
  - Dr R Dulabh, Johannesburg, Gauteng
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Roodepoort Medicross Clinical Research Centre, Roodepoort, Gauteng
  - Dr Pillay's Rooms, Durban, KwaZulu-Natal
  - Clinical Research Institute of South Africa, KwaDukuza, KwaZulu-Natal
  - Langeberg Clinical Trials, Cape Town, Western Cape
- Turkey (Türkiye) (4):
  - Akdeniz University Tip Fakultesi Hastanesi, Antalya
  - Seyrantepe Hamidiye Etfal Egitim ve Arastirma Hastanesi, Istanbul
  - T.C. Saglik Bakanligi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Tekirdag Namık Kemal UTF, Tekirdağ

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com